CLINICAL TRIAL: NCT01324440
Title: A Randomized, Multicenter, Double-Blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Single Dose of Merck 0657nI Staphylococcus Aureus Vaccine With Merck Aluminum Adjuvant or Without Merck Aluminum Adjuvant in Healthy Adults 18 to 70 Years of Age
Brief Title: Safety, Tolerability, and Immunogenicity of a Single Dose of Merck 0657nI Staphylococcus Aureus Vaccine With or Without Merck Aluminum Adjuvant (V710-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V710-002
Record Dates: First submitted 2011-02-24; First posted 2011-03-29 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Staphylococcal Infections
Keywords: Bacterial Vaccines; Staphylococcus Aureus; Adjuvanted Vaccine
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- V710 without MAA (Experimental)
  Interventions: Biological: V710 (30 µg) without MAA
- V710 with MAA (Active Comparator)
  Interventions: Biological: V710 (30 µg) with MAA

INTERVENTIONS:
Biological: V710 (30 µg) with MAA — Single 0.5-mL injection (30-µg) of V710 with MAA, intramuscularly
  Arms: V710 with MAA
Biological: V710 (30 µg) without MAA — Single 0.5-mL injection (30-µg) dose of V710 without MAA, intramuscularly
  Arms: V710 without MAA

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and immunogenicity of the Merck 0657nI S. aureus vaccine (V710) either with or without Merck Aluminum Adjuvant (MAA).

ELIGIBILITY:
Inclusion criteria:

* Participant was in good physical health
* Participant was able to understand study procedures and agreed to participate in the study by providing written informed consent.
* Participant was willing and able to participate in the entire study duration planned for up to 12 months (~360 days).
* Female participants of reproductive potential were required to have a negative urine pregnancy test immediately prior to study vaccination. Female participants of reproductive potential must have used an acceptable method of birth control for 2 weeks prior to enrollment, and agreed to use an acceptable method of birth control for 1 month after vaccination.

Exclusion criteria:

* Participant suffered from a chronic skin condition that predisposed the individual to the development of chronic skin or soft-tissue infections (e.g., psoriasis, chronic granulomatous disease, atopic dermatitis).
* Participant developed a serious infection (e.g., bacteremia, pneumonia, mediastinitis) attributed to S. aureus in the 12 months prior to screening.
* Participant had a history of anaphylaxis to aluminum-containing adjuvant or other vaccine components.
* Participant had a temperature of ≥100.4ºF (≥38.0ºC), oral equivalent, within 48 hours prior to receipt of V710.
* Participant had received a live virus vaccine within 30 days prior to receipt of V710 or was scheduled to receive vaccination with a live virus vaccine within 30 days following study entry.
* Participant had received any other licensed vaccine (including non-live virus vaccines) within 14 days prior to receipt of V710 or was scheduled to receive any other licensed vaccine (including non-live virus vaccines) within 30 days following study entry.
* Participant had received V710 in a prior clinical study (Merck V710 Protocol 001).
* Participant was administered immunoglobulin or blood product within 90 days prior to receipt of V710 or was scheduled to receive such products within 30 days following study entry.
* Participant had received treatment with systemic (intramuscular, oral, or intravenous) corticosteroids or another immunosuppressive medication (e.g., calcineurin inhibitors, mycophenolate, azathioprine) or biological agents (e.g., rituximab) in the 14 days prior to receipt of V710 or was anticipated to receive such medications for a chronic medical condition during the course of the study.
* Participant had a condition that required active medical intervention or monitoring to avert serious danger to the participant's health or well-being, such as diabetes mellitus, autoimmune disease, or clinically significant chronic medical conditions that were considered progressive, including but not limited to: coronary artery disease, congestive heart failure, cardiomyopathy, progressive valvular heart disease, chronic obstructive pulmonary disease, pulmonary fibrosis, active peptic ulcer disease, chronic renal disease, chronic hepatic disease, multiple sclerosis, progressive neuropathies, or seizure disorder requiring therapy in the past 3 years.
* Participant had known or suspected impairment of immunologic function including, but not limited to, the following conditions: autoimmune disease, diabetes mellitus, endstage renal disease, hepatic insufficiency/cirrhosis, splenectomy, or human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS).
* Participant had a condition in which repeated venipuncture or injections posed more than minimal risk for the subject, such as hemophilia, other severe coagulation disorders, or significantly impaired venous access.
* Participant was pregnant or breastfeeding, or planning to conceive within the 12-month study duration period.
* Participant had clinically significant abnormalities based on the participant or physical examination.
* Participant had recent history (within the past 5 years) or current evidence of drug or alcohol abuse.
* Participant had a major psychiatric illness, including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, or any subject with suicidal ideation within the previous 3 years.
* Participant was legally or mentally incapacitated.
* Participant had participated in another clinical study in the past 4 weeks, or participant planned to participate in a treatment-based study or study in which an invasive procedure was to be performed during the first 3 months of this study (through Day 84).
* Participant had a history of any condition which, in the opinion of the investigator, posed an additional risk for the subject or confounded the results of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

REFERENCES:
- [Result] Harro CD, Betts RF, Hartzel JS, Onorato MT, Lipka J, Smugar SS, Kartsonis NA. The immunogenicity and safety of different formulations of a novel Staphylococcus aureus vaccine (V710): results of two Phase I studies. Vaccine. 2012 Feb 21;30(9):1729-36. doi: 10.1016/j.vaccine.2011.12.045. Epub 2011 Dec 20. PMID 22192849

RESULTS

PARTICIPANT FLOW:
Groups:
- V710 With MAA: Single 0.5-mL injection (30-µg) dose of V710 with MAA, intramuscularly.
- V710 Without MAA: Single 0.5-mL injection (30-µg) dose of V710 without MAA, intramuscularly.
Period: Overall Study
Arm/Group | V710 With MAA | V710 Without MAA
Started | 32 | 32
Completed | 32 | 31
Not Completed | 0 | 1
Not completed — Subject moved | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V710 With MAA | V710 Without MAA | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Customized [Number; unit: participants]
  17 and under | 0 | 0 | 0
  18 to 29 | 6 | 5 | 11
  30 to 39 | 1 | 4 | 5
  40 to 49 | 9 | 7 | 16
  50 to 59 | 12 | 10 | 22
  60 to 69 | 4 | 6 | 10
  Over 69 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Immune Response, Defined as a Change in Antibody Level Greater Than or Equal to a 2-fold-rise at Day 14 Compared to Baseline
Description: Immunoglobulin G (IgG) antibodies were measured by a LUMINEX(TM) assay.
Time Frame: Baseline and Day 14 postvaccination
Population: The per-protocol analysis excluded patients who had missing baseline and/or postvaccination (Day 14) serology data and patients who developed a S. aureus infection during the 14 days postvaccination.
Measure: Number; unit: participants
Arm/Group | V710 With MAA | V710 Without MAA
Number analyzed (Participants) | 32 | 32
participants | 27 | 23

2. Primary Outcome: Geometric Mean Antibody Concentrations (GMC)
Description: Immunoglobulin G (IgG) antibodies were measured by a LUMINEX(TM) assay.
Time Frame: Day 14 postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | V710 With MAA | V710 Without MAA
Number analyzed (Participants) | 32 | 32
mcg/mL | 115.4 [82.9 to 160.6] | 99.1 [73.5 to 133.6]

3. Primary Outcome: Change in Antibody Concentration (Titer) at Day 14 Compared to Baseline, Expressed as the Geometric Mean Fold-rise (GMFR)
Description: Immunoglobulin G (IgG) antibodies were measured by a LUMINEX(TM) assay.
  The GMFR is the ratio of the antibody concentration at Day 14 to the antibody concentration at baseline.
Time Frame: Baseline and Day 14 postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of IgG titer at Day 14 to baseline
Arm/Group | V710 With MAA | V710 Without MAA
Number analyzed (Participants) | 32 | 32
ratio of IgG titer at Day 14 to baseline | 4.5 [3.3 to 6.1] | 4.0 [2.9 to 5.4]

4. Primary Outcome: Number of Vaccine-related Serious Adverse Experiences
Description: Investigators were instructed to determine the seriousness and causality (relatedness to test vaccine) of each AE based on criteria defined in the protocol:
  A serious adverse event (SAE) is any AE that:
  * results in death,
  * is life threatening,
  * results in a persistent or significant disability/incapacity,
  * results in or prolongs an existing inpatient hospitalization,
  * is a congenital anomaly/birth defect,
  * is a cancer,
  * is an overdose,
  * or is another important medical event that may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to Day 360 postvaccination
Population: Any subject who received clinical material and had at least 1 day of safety follow-up was included in the safety summary.
Measure: Number; unit: participants
Arm/Group | V710 With MAA | V710 Without MAA
Number analyzed (Participants) | 32 | 32
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | V710 With MAA | V710 Without MAA
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 21/32 | 17/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V710 With MAA (N=32) | V710 Without MAA (N=32)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (3)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 3 (3) | 1 (1)
Injection site erythema (General disorders) | 4 (4) | 2 (2)
Injection site pain (General disorders) | 10 (11) | 6 (8)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 2 (2) | 4 (4)
Injection site warmth (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 6 (6)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.